CLINICAL TRIAL: NCT07074613
Title: The Effects of Augmented Reality Treadmill Walking on Cognitive Function, Body Composition, Physiological Responses, and Acceptability in Older Adults: A Randomized Controlled Trial
Brief Title: Augmented Reality Treadmill Walking for Cognitive and Physical Health in Older Adults
Acronym: ART-Walk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan College of Performing Arts (Other)
Responsible Party: Principal Investigator, CHENG-EN WU, Assistant Professor, Office of Physical Education, National Taiwan College of Performing Arts
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114-86; IRB No. 114-86 (Other: City Hospital Renai IRB)
Record Dates: First submitted 2025-06-26; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Aging; Cognitive Decline; Sarcopenia; Mobility Limitation; Balance Impairment
Keywords: Augmented Reality; Treadmill Walking; Older Adults; Cognitive Function; Body Composition; Balance Training; Sarcopenia Intervention; Technology Acceptance; Physical Activity; Gait Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Sarcopenia; Mobility Limitation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: an experimental group that received augmented reality treadmill walking training and a control group that received traditional treadmill walking training. Both groups participated in the same frequency and duration of exercise (3 sessions per week for 12 weeks), allowing direct comparison of intervention effects on cognitive function, body composition, and physiological responses.
Masking Description: No masking was used in this study. Due to the nature of the intervention (visible augmented reality equipment), participants, investigators, and outcome assessors were aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Augmented Reality Treadmill Walking (Experimental): Participants in this group performed treadmill walking using the JOHNSON 8.1T treadmill with Passport AR system. The device provided immersive visual environments (e.g., forest trails, hills) and real-time feedback on heart rate, speed, and distance.
  Each participant completed supervised walking sessions 3 times per week for 12 weeks, with each session lasting 60 minutes (10-minute warm-up, 40-minute walking, 10-minute cool-down).
  Interventions: Device: JOHNSON 8.1T treadmill with Passport AR system
- Active Comparator: Traditional Treadmill Walking (Active Comparator): Participants in this group performed treadmill walking using the CHANSON CS-6630 treadmill, which provided standard speed, time, and distance tracking without augmented reality features.
  Each participant completed supervised walking sessions 3 times per week for 12 weeks, with each session lasting 60 minutes (10-minute warm-up, 40-minute walking, 10-minute cool-down).
  Interventions: Device: Traditional Treadmill Walking

INTERVENTIONS:
Device: Traditional Treadmill Walking — Participants walked on a traditional treadmill with standard time, speed, and distance tracking, no AR features.
  Other Names: CHANSON CS-6630 treadmill
  Arms: Active Comparator: Traditional Treadmill Walking
Device: JOHNSON 8.1T treadmill with Passport AR system — Participants walked on an AR-integrated treadmill with immersive virtual environments and real-time feedback.
  Arms: Experimental: Augmented Reality Treadmill Walking

SUMMARY:
This study evaluated the feasibility and health effects of using augmented reality (AR) treadmill walking in older adults. Sixty community-dwelling adults aged 65 to 80 years were randomly assigned to either an AR treadmill group or a traditional treadmill group. Both groups participated in supervised walking sessions three times per week for twelve weeks. The study examined changes in mobility, balance, body composition, physiological responses, and participants' perceptions of the AR technology.

DETAILED DESCRIPTION:
This randomized controlled trial evaluated the effects of augmented reality (AR) treadmill walking on mobility-related motor function, body composition, physiological responses, and technology acceptance among older adults. A total of 60 community-dwelling adults aged 65 to 80 years were randomly assigned to either an experimental group (AR treadmill walking) or a control group (traditional treadmill walking).

Participants in both groups engaged in supervised walking sessions three times per week for twelve weeks. Each session lasted 60 minutes, including a 10-minute warm-up, 40-minute treadmill walking, and a 10-minute cool-down. The AR treadmill (JOHNSON 8.1T) provided immersive visual environments and real-time feedback on physiological data. The control group used a standard treadmill (CHANSON CS-6630) without AR features.

Primary outcome measures included stride length, gait speed, and balance. Secondary outcomes included skeletal muscle mass, body fat mass, body fat percentage, heart rate, calorie expenditure, walking distance, and technology acceptance assessed by a validated questionnaire.

Statistical analysis included repeated-measures ANOVA, independent t-tests, and Pearson correlation analysis to examine group differences and associations between physiological responses and technology acceptance.

ELIGIBILITY:
Inclusion Criteria:

Community-dwelling adults aged 65 to 80 years

Able to walk independently without assistive devices

Cognitively intact and able to follow instructions

No prior use of augmented reality (AR) exercise programs within the past 3 months

Willing to participate in the study and provide informed consent

Exclusion Criteria:

Diagnosed with chronic conditions that impair mobility (e.g., cardiovascular disease, severe arthritis)

Severe visual or auditory impairments that affect interaction with AR equipment

Neurological or psychiatric disorders that may interfere with participation

Known susceptibility to motion sickness or discomfort with virtual environments (AR-induced discomfort)

Inability to complete the 12-week training protocol or attend scheduled assessments

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Stride Length | Baseline and after 12 weeks of intervention
  Average stride length (in centimeters) measured using the 2-Minute Walk Test (2MWT).
Gait Speed | Baseline and after 12 weeks of intervention
  Walking speed (in meters per second) assessed during a 30-meter walk test.
Balance (Timed Up and Go Test) | Baseline and after 12 weeks of intervention
  Time taken to complete the Timed Up and Go (TUG) test. Lower values indicate better balance.

SECONDARY OUTCOMES:
Skeletal Muscle Mass | Baseline and after 12 weeks of intervention
  Measured using bioelectrical impedance analysis (InBody 520). Unit: kg.
Body Fat Mass | Baseline and after 12 weeks of intervention
  Measured using bioelectrical impedance analysis (InBody 520). Unit: kg.
Body Fat Percentage | Baseline and after 12 weeks of intervention
  Measured using bioelectrical impedance analysis (InBody 520). Unit: %.
Heart Rate | During each session (12 weeks)
  Average heart rate monitored during each exercise session using treadmill sensors or wearable device.
Calorie Expenditure | During each session (12 weeks)
  Calories burned per session, tracked by treadmill and validated device.
Distance Walked | During each session (12 weeks)
  Total distance covered per session (in meters or kilometers).
Technology Acceptance | After 12 weeks of intervention
  Measured using a validated questionnaire based on the Technology Acceptance Model (TAM), including perceived ease of use, usefulness, and behavioral intention.

CONTACTS AND LOCATIONS:
Locations (1):
- Fitness Center, National Taiwan College of Performing Arts, Taipei, No. 177, Section 2, Neihu Rd., Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy considerations and the small sample size of older adult participants. Additionally, data sharing was not included in the original study protocol or informed consent process. Therefore, public sharing of IPD is not permitted under the current ethical approval.

DOCUMENTS (1):
  • Informed Consent Form (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT07074613/ICF_000.pdf